CLINICAL TRIAL: NCT07113067
Title: Accelerated rTMS for Post-stroke Apathy: A Double-blind Randomized Controlled Trial
Brief Title: Accelerated rTMS vs. Sham for Stroke Apathy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00144684
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Apathy; Stroke; Stroke Sequelae; Stroke/Brain Attack; Stroke/ Cerebrovascular Accident (Ischemic or Hemorrhagic); Motivation; Abulia
Keywords: Depression; Stroke; Stroke Recovery; Apathy; TMS; Motivation; Abulia; Amotivation
MeSH Terms: conditions — Lethargy; Stroke; Ischemia; Depression | interventions — Transcranial Magnetic Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants and members of the research team except for the statistician will be blinded as to which arm participants are in until the conclusion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): This group will receive active accelereated iTBS-rTMS
  Interventions: Device: MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System (Active); Other: Brainsight Neuronavigation System
- Sham TMS (Sham Comparator): This group will receive sham accelerated iTBS-rTMS
  Interventions: Device: MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System (Sham); Other: Brainsight Neuronavigation System

INTERVENTIONS:
Device: MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System (Active) — Active treatment will consist of high-dose iTBS-rTMS to left dmPFC delivered in runs of 600 pulses at an intensity of 120% resting motor threshold (rMT). iTBS triplets at 50 Hz will be delivered for 2 seconds, repeated every 10 seconds for a total of 190 seconds. Each session will be separated by at least 10-15 minutes and a total of 12 sessions will be given on each treatment day (3-4 hours per study day). A total of 43,200 pulses will be delivered over the entire six days of treatment.
  Other Names: Active TMS
  Arms: Active TMS
Device: MagVenture MagPro Transcranial Magnetic Stimulation (TMS) System (Sham) — For the sham stimulation group, a focal electric sham will be used which is indistinguishable from active TMS including a pretreatment individualized sham titration, sham outputs noises synchronized to pulse delivery, and an individualized level of sham stimulation throughout the treatment.
  Technicians administering active vs sham TMS will be masked by using a random code generated by the statistician that will indicate whether to use the active or sham side of the coil. Treatments will appear identical to the technician regardless of whether active or sham TMS is administered.
  Other Names: Sham TMS
  Arms: Sham TMS
Other: Brainsight Neuronavigation System — A brainsight neuronavigation system will be used during TMS treatments to target treatment location using individual MRI data

SUMMARY:
Apathy is a common set of symptoms seen in many people following a stroke. Apathy occurs when a person has lost motivation, becomes withdrawn, and stops doing things that used to be important to them. Apathy has a large negative impact on a person's quality of life, and can also have a large impact the people who take care of them. There are currently no FDA-approved treatments to help with apathy, and other services like therapy may be difficult to access for people who have had a stroke. To address this problem, investigators are conducting a study to find out if a form of treatment called repetitive transcranial magnetic stimulation (rTMS) can be safe and helpful for people struggling with apathy after a stroke. This study will apply a new form of rTMS which can be delivered quickly to a part of the brain called the medial prefrontal cortex (mPFC). This study will help establish whether this treatment is safe, comfortable, and effective for people with apathy after a stroke, and will help researchers develop new forms of treatment.

DETAILED DESCRIPTION:
Apathy is a significant source of disability in a wide range of neurodegenerative conditions, including prominently in stroke (40-60% of stroke survivors). Furthermore, the amotivation that characterizes apathy fundamentally interferes with quality of life and specifically with rehabilitation. At the extreme, it has been associated with post-stroke suicide risk.

Notably, previous research has demonstrated that apathy is distinct from post-stroke depression, fatigue, and other affective and cognitive impairments and often persists despite improvements in these associated domains. Existing literature has implicated the anterior cingulate cortex (ACC) in transdiagnostic amotivation and apathy. The dorsal medial prefrontal cortex (dmPFC) lies immediately superficial to the ACC and, via strong functional and structural interconnections and, makes this a promising target for repetitive transcranial magnetic stimulation (rTMS) to modify the substrates of apathy and is a safe and acceptable stimulation target.

Furthermore, rTMS is especially promising for post-stroke apathy (PSA) as it provides the flexibility for personalizing TMS coil placement in relation to post-stroke brain network anomalies, which vary significantly across stroke survivors. A typical course of rTMS entails one treatment/day for 4 to 6 weeks (30-40 sessions), which can be burdensome and reduce adherence, particularly for those with mobility limitations, as is common in stroke. Accelerated rTMS, a recent innovation in which multiple sessions are delivered each day to reduce treatment burden, is safe and effective in depression.

As a first test of suitability in post-stroke apathy (n=14), investigators conducted an open-label pilot trial that delivered 12 sessions of 600 pulses of accelerated intermittent theta burst (iTBS)-rTMS on each of three days within one week to dmPFC (36 total sessions; 21,600 total pulses). Targeting was standardized using neuronavigation and MNI coordinates to position the TMS coil over the left dmPFC. No adverse neuroradiological, neurocognitive, or neuropsychiatric effects were noted coupled with high retention (>80%) and acceptability ratings. Furthermore, while this Phase I pilot trial was not dosed for efficacy, investigators observed significant effect size (Cohen's d on the Lille Apathy Rating Scale from baseline to one-month was 0.61 along with improvements in apathy, improved quality of life with reduced caregiver burden.

In a separate ongoing dose-response study in the MUSC Brain Stimulation Lab, accelerated iTBS to left dlPFC was applied for up to 10 sessions per day for 5 days, maximum 50 active sessions, 30,000 individual total pulses among individuals with moderate to severe anxiety and depression. The preliminary findings suggest that psychosocial functioning/quality of life improves at higher doses, and the emerging dose-response curve suggests the asymptote is likely above the maximum dose tested (i.e., 10 sessions/day).

Taken together, 1) accelerated rTMS is safe and effective, 2) has the potential to rapidly remediate cross-domain neuropsychiatric impairment in chronic stroke, including apathy and 3) examining higher dose is warranted to optimize outcomes.

In this present study we will examine 1) the efficacy of active relative to sham stimulation in a double-blind, randomized design, 2) safety, acceptability, and efficacy of higher dosing in stroke patients 3) durability, 4) generalizability of gains in other neuropsychiatric and neurocognitive domains outside apathy.

Specifically, we will conduct a double-blind, randomized, sham controlled phase I/II trial of accelerated iTBS-rTMS for PSA and associated impairments in chronic stroke. 36 patients (age 40-80 years) with PSA secondary to ischemic or hemorrhagic stroke (≥6 months chronicity) will be recruited and randomized 1:1 to two stimulation groups: 1) active iTBS to left dmPFC targeted to standardized MNI coordinates, or 2) electrical sham.

Protocol, target location, and assessments will mirror our Phase 1 trial, in which investigators observed large open-label effects, except in this study, investigators will increase to 6 days of treatment over 2 weeks (total 72 sessions; 43,200 total pulses), enabling assessment of efficacy and durability over follow-up.

Participants will undergo clinical assessments at baseline, immediately post-treatment, and 1-month follow-up. Brain MRIs will be collected at pre- and immediately post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or greater
* Right- or left-hemisphere ischemic or hemorrhagic stroke with at least 6 months chronicity
* Symptomatic apathy as confirmed by (A) total score on the Apathy Evaluation Scale by the participant or the caregiver/co-participant (AES) of ≥39
* Ability to participate in psychometric testing and cognitive tasks
* Intact cortex at the TMS target site as confirmed by pre-treatment MRI
* Ability to have a co-participant/caregiver who meets the criteria as detailed below.

Exclusion Criteria:

* Primary extra-axial hemorrhage (subdural or subarachnoid) without ischemic stroke or intraparenchymal hemorrhage
* Concomitant neurological disorders affecting motor or cognitive function (e.g. dementia)
* Moderate or severe global aphasia
* Visual impairment precluding completion of cognitive tasks
* Presence of contraindications to MRI or TMS including electrically, magnetically or mechanically activated metal or nonmetal implants such as cardiac pacemaker, intracerebral vascular clips or any other electrically sensitive support system;
* Pregnancy (to be later confirmed by UPT in any premenopausal female participants)
* History of a seizure disorder
* Preexisting scalp lesion, wound, bone defect, or hemicraniectomy
* Claustrophobia precluding ability to undergo an MRI
* Active substance use disorder
* Psychotic disorders
* Bipolar 1 Disorder
* Acute suicidality as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)30 or suicide attempt in the previous year

For CO-PARTICIPANT/CAREGIVER:

Inclusion Criteria:

* Age 18 years or older
* Is a reliable informant who has at least weekly contact with the participant and can speak to the participant's cognitive and everyday functioning.

Exclusion Criteria:

- Unable to engage with study procedures in which Co-Participant input is needed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in apathy symptoms, as measured by the Lille Apathy Rating Scale (LARS) compared to baseline | Pre-treatment, immediately post-treatment, and at one month post-treatment follow-up
  The Lille Apathy Rating Scale (LARS) is a clinically validated 33-item structured interview assessing clinical symptoms of apathy. The structured interview is broken into 9 sub-scales including everyday productivity, interests, taking the initiative, novelty seeking, motivation, emotional responsiveness, concern, and social life. Total scores can range from -36 to +36 and are further stratified by factorial sub-scores including intellectual curiosity, emotion, action initiation, and self-awareness.
Change in apathy symptoms as measured by the Apathy Evaluation Scale (AES) - Self and Informant Versions | Pre-treatment, immediately post-treatment, and weekly for four weeks post-treatment.
  The Apathy Evaluation Scale (AES) clinically validated rating scale assessing symptoms of apathy. The AES is comprised of 18 items rated on a four-point Likert-Scale assessing and quantifying emotional, behavioural and cognitive aspects of apathy. Total scores on the AES range from 18 to 72 with high scores correlating with greater severity of apathy.
Incidence of Treatment-Emergent Adverse Events and Side Effects as assessed by change in the Review of Systems Criteria compared to baseline | After each session of rTMS during each of six treatment days within two weeks
  A review of systems questionnaire will be administered to rate the subjective symptom (headache, scalp pain, arm/hand pain, other pain(s), numbness/tingling, other sensation(s), weakness, loss of dexterity, vision/hearing change(s), ear ringing, nausea/vomiting, appetite loss, rash, skin change(s) or any other symptom(s)) on a scale of 0 to 5 (none, minimal, mild, moderate, marked, severe).
Change From Baseline Cognition, as Measured by the Fluid Cognition Composite Score From the NIH Toolbox Cognition Battery compared to baseline | Pre-treatment, immediately post-treatmen
  Fluid cognition was measured using the iPad-administered NIH Toolbox Cognition Battery (NIHTB-CB). Fluid Cognition Composite scores were calculated by averaging the demographically adjusted (age, education, sex, race/ethnicity; Casaletto et al., 2015) T-scores for 4 NIHTB-CB tests: the flanker inhibitory control, list sorting working memory, pattern comparison processing speed, and dimensional change card sort tests. T-Scores have a mean of 50 and a standard deviation of 10. Lower scores indicate worse performance.
Participant retention rate | calculated at the end of the study follow-up assessment period (one month post-treatment)
  Percentage of participants who completed the study relative to all participants who initiated treatment. Percentage of participants who completed the study relative to all participants who initiated treatment. Percentage of participants who completed the study relative to all participants who initiated treatment.
Patient perception of treatment acceptability as assessed by study-specific questionnaire | After each session of rTMS during each of three treatment days within one week, and at one month post-treatment follow-up
  A 15-item study-specific questionnaire of rTMS treatment acceptability, with each item rated on a scale from 1 to 5 (1 = not at all, 3 = somewhat, 5 = very much so). Higher scores indicate better acceptability for the first 10 items, lower scores indicate better acceptability for the last 5 items.
Frontal Systems Behavior Scale (FrSBE)-Apathy scale | Pre-treatment, post-treatment and at 4 weeks post treatment
  The Frontal Systems Behavior Scale (FrSBE) assesses behavioral changes associated with frontal lobe dysfunction, including apathy, disinhibition, and executive deficits. In this study, apathy-as measured by the FrSBE Apathy subscale-is the primary outcome.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form | Pre-treatment, immediately post-treatment, and weekly for four weeks post-treatment
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form The Patient-Reported Outcomes Measurement Information System (PROMIS) is a clinically validated adaptive clinical assessment tool designed under the NIH to capture patient-reported symptoms in several psychiatric symptom domains for use in clinical research.

CONTACTS AND LOCATIONS:
Overall Officials: Parneet Grewal, PhD, Principal Investigator — Medical University of South Carolina; Lisa McTeague, PhD, Principal Investigator — Medical University of South Carolina; Kevin Caulfield, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Brain Stimulation Lab, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared in publications, ClinicalTrials.gov, or data repositories.

REFERENCES:
- [Background] Marin RS, Biedrzycki RC, Firinciogullari S. Reliability and validity of the Apathy Evaluation Scale. Psychiatry Res. 1991 Aug;38(2):143-62. doi: 10.1016/0165-1781(91)90040-v. PMID 1754629
- [Background] Casaletto KB, Umlauf A, Beaumont J, Gershon R, Slotkin J, Akshoomoff N, Heaton RK. Demographically Corrected Normative Standards for the English Version of the NIH Toolbox Cognition Battery. J Int Neuropsychol Soc. 2015 May;21(5):378-91. doi: 10.1017/S1355617715000351. Epub 2015 Jun 1. PMID 26030001
- [Background] Sockeel P, Dujardin K, Devos D, Deneve C, Destee A, Defebvre L. The Lille apathy rating scale (LARS), a new instrument for detecting and quantifying apathy: validation in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2006 May;77(5):579-84. doi: 10.1136/jnnp.2005.075929. PMID 16614016
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Levy R, Dubois B. Apathy and the functional anatomy of the prefrontal cortex-basal ganglia circuits. Cereb Cortex. 2006 Jul;16(7):916-28. doi: 10.1093/cercor/bhj043. Epub 2005 Oct 5. PMID 16207933
- [Background] Jorge RE, Starkstein SE, Robinson RG. Apathy following stroke. Can J Psychiatry. 2010 Jun;55(6):350-4. doi: 10.1177/070674371005500603. PMID 20540829
- [Background] Santa N, Sugimori H, Kusuda K, Yamashita Y, Ibayashi S, Iida M. Apathy and functional recovery following first-ever stroke. Int J Rehabil Res. 2008 Dec;31(4):321-6. doi: 10.1097/MRR.0b013e3282fc0f0e. PMID 19008681
- [Background] Le Heron C, Apps MAJ, Husain M. The anatomy of apathy: A neurocognitive framework for amotivated behaviour. Neuropsychologia. 2018 Sep;118(Pt B):54-67. doi: 10.1016/j.neuropsychologia.2017.07.003. Epub 2017 Jul 8. PMID 28689673
- [Background] Sasaki N, Hara T, Yamada N, Niimi M, Kakuda W, Abo M. The Efficacy of High-Frequency Repetitive Transcranial Magnetic Stimulation for Improving Apathy in Chronic Stroke Patients. Eur Neurol. 2017;78(1-2):28-32. doi: 10.1159/000477440. Epub 2017 Jun 3. PMID 28578330
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360